CLINICAL TRIAL: NCT02870907
Title: Adjuvant Treatment in Extensive Unilateral Retinoblastoma Primary Enucleated
Brief Title: Adjuvant Treatment in Extensive Unilateral Retinoblastoma Primary Enucleated (RB SFCE 2009)
Acronym: RB SFCE 09
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2009-04
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Retinoblastoma
Keywords: primary enucleation; retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Observation; Etoposide; Vincristine; Carboplatin; Cyclophosphamide; Thiotepa; Cytapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low risk group (Experimental): No treatment
  Interventions: Other: Observation
- Intermediate risk sub group 1 (Experimental): 2 cycles (4 courses): 2 courses of etoposide and Carboplatin from D1 to D5 and Vincristin at D22 and D26- Cyclophosphamide from D22 to D26.
  Interventions: Drug: Etoposide; Drug: Carboplatin; Drug: Vincristine; Drug: Cyclophosphamide
- Intermediate risk sub group 2 (Experimental): 2 courses of Vincristin and Carboplatin
  Interventions: Drug: Vincristine; Drug: Carboplatin
- High risk group (Experimental): * Orbital irradiation
  * 3 cycles of two different types of alternating chemotherapy courses (id 6 courses) :
    * Etoposide (100 mg/m²/d) and Carboplatin (160 mg/m²/d) with intrathecal Thiotepa injection.
    * Vincristin (1,5 mg/m²/d) - Cyclophosphamide (1000 mg/m²/d)
    * Cytapheresis for peripheral blood stem cells collection after the primary or the secondary courses of Vincristine- Cyclophosphamide.
  * High dose chemotherapy :
    * Carboplatin (AUC : 7/d) - etoposide (250 mg/m²/d) - Thiotepa (300 mg/m²/d)
    * Peripheral bood stem cell transplantation.
  Interventions: Radiation: Orbital irradiation; Drug: Etoposide; Drug: Carboplatin; Drug: Thiotepa; Drug: Vincristine; Drug: Cyclophosphamide; Procedure: Cytapheresis; Procedure: Peripheral bood stem cell transplantation

INTERVENTIONS:
Other: Observation — no post operative chemotherapy
  Other Names: Low risk group
  Arms: Low risk group
Drug: Etoposide — 100 mg/m²/d, IV (in the vein) from D1 to D5.
  Other Names: Intermediate risk sub group 1
  Arms: Intermediate risk sub group 1
Drug: Vincristine — 1, 5 mg/m²/d, IV at D1.
  Other Names: Intermediate risk sub group 2
  Arms: Intermediate risk sub group 2
Radiation: Orbital irradiation — 45 Grays (Standard or external beam radiotherapy).
  Other Names: High risk group
  Arms: High risk group
Drug: Carboplatin — 160 mg/m²/d, IV from D1 to D5.
  Other Names: Intermediate risk sub group 1
  Arms: Intermediate risk sub group 1
Drug: Vincristine — 1,5 mg/m²/d, IV at D22 and D26
  Other Names: Intermediate risk sub group 1
  Arms: Intermediate risk sub group 1
Drug: Cyclophosphamide — 300 mg/m²/d, IV from D22 to D26.
  Other Names: Intermediate risk sub group 1
  Arms: Intermediate risk sub group 1
Drug: Carboplatin — 560 mg/m²/d, IV at D1.
  Other Names: Intermediate risk sub group 2
  Arms: Intermediate risk sub group 2
Drug: Etoposide — 100 mg/m²/d, IV from D1 to D5
  Other Names: High risk group
  Arms: High risk group
Drug: Carboplatin — 160 mg/m²/d,IV from D1 to D5
  Other Names: High risk group
  Arms: High risk group
Drug: Thiotepa — 15 mg, intrathecal Thiotepa injection at D1.
  Other Names: High risk group
  Arms: High risk group
Drug: Vincristine — 1,5 mg/m²/d), IV at D22
  Other Names: High risk group
  Arms: High risk group
Drug: Cyclophosphamide — 1000 mg/m²/d, IV from D22 à D24.
  Other Names: High risk group
  Arms: High risk group
Procedure: Cytapheresis — Cytapheresis for peripheral blood stem cells collection after the primary or the secondary courses of Vincristine- Cyclophosphamid.
  Other Names: High risk group
  Arms: High risk group
Drug: Carboplatin — AUC : 7/d, IV from D-8 to D-6.
  Other Names: High risk group
  Arms: High risk group
Drug: Etoposide — 250 mg/m²/d, IV from D -5 to D-3.
  Other Names: High risk group
  Arms: High risk group
Drug: Thiotepa — 300 mg/m²/d, IV from D-5 to D-3.
  Other Names: High risk group
  Arms: High risk group
Procedure: Peripheral bood stem cell transplantation — at D0
  Other Names: High risk group
  Arms: High risk group

SUMMARY:
Postoperative Treatment of Unilateral Retinoblastoma After Primary Enucleation according to histopathological risk factors of the International Retinoblastoma Staging Working Group.

DETAILED DESCRIPTION:
Post operative chemotherapy +/- radiotherapy according to histopathological risk factors of the International Retinoblastoma Staging Working Group.

* Low risk group :

  * No optic nerve involvement.
  * Intra and prelaminar involvement
  * No choroidal involvement.
  * Minimal superficial choroidal involvement .
* Intermediate risk group, 2 sub groups :

  * Sub group 1 :

    * Retrolaminar involvement without Invasion of surgical margin associated or not to massive choroidal involvement
    * Anterior segment involvement.
    * Intrascleral involvement.
  * Sub Group 2 :

    * Isolated massive choroidal involvement.
* High risk group :

  * Invasion of the surgical margin of the optic nerve
  * and/or microscopic extrascleral involvement
  * Optic nerve meningeal sheat involvement .

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent - a signed informed consent and/or assent (as age appropriate) will be obtained according to institutional guidelines;
2. Male or female ≥2 months and <10 years of age at the time of signing the informed consent form;
3. Diagnosis of non familial extensive unilateral retinoblastoma treated by primary enucleation
4. In case of post operative chemotherapy, patients must have adequate organ function:

   * Adequate hematopoietic function Neutrophils>1.0x109/l, Platelets >100 x 109/l.
   * Adequate hepatic function: grade II NCI CTC
   * Adequate renal function: serum creatinemia <1.5 x ULN for age with normal creatinine clearance estimated by SCHWARTZ formula
   * Audiometry < Grade II de Brock.
   * Echocardiography normal in case of high dose cyclophosphamide chemotherapy (3 g/m²).
5. Patients affiliated to a Social Security Regimen or beneficiary of the same
6. No chemotherapy or radiotherapy prior to administration of the first dose of study treatment for retinoblastoma or other tumor types
7. Without medical cons-indication to study drugs.

Exclusion Criteria:

* Bilateral and/or familial or trilateral retinoblastoma.
* Unilateral retinoblastoma with indication of primary chemotherapy before enucleation:

  * One or several surgical risk factors
  * Buphthalmia Exophthalmia.
  * Peri ocular inflammatory signs.
  * Extraocular extension :
  * Radiological retrolaminar extension (more than 3 mm behind the lamina cribrosa) and or meningeal sheat optic nerve extension.
  * Extrascleral extension
  * Lymp nodes extension
* Unilateral retinoblastoma with possibility of conservative treatment:
* Metastatic extension at diagnosis
* One inclusion criteria non observed
* Uncontrolled medical conditions, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2010-03-18 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of extra ocular relapses | 5 years

SECONDARY OUTCOMES:
Evaluate long term and acute toxicities of adjuvant chemotherapy and orbital irradiation if necessary. | 5 years
  Number of participants with treatment-related Adverse Events as assessed by CTCAE v3.0.
Number of patient with secondary bilateralisation | 5 years
Evaluate the different histopathological risk factors frequency | 5 years
  Number of patient in each histopathological risk group
To determine tumors genomic | at the inclusion
  Tumor genomic characterization in order to provide some new prognosis factors and better understanding of tumorigenesis by using of NGS (Next Generation Sequencing) techniques
Evaluate sensitivity of MRI in detecting extra ocular extension | At the inclusion
  Number of extra ocular extension detected by MRI

CONTACTS AND LOCATIONS:
Locations (27):
- France (27):
  - Chr Felix Guyon, Saint-Denis, La Réunion
  - Hopital Nord Chu Amiens, Amiens
  - Chu Angers, Angers
  - Hopital Jean Minioz, Besançon
  - Chu R; Pellegrin, Bordeaux
  - Chu Morvan, Brest
  - CHU CAEN, Caen
  - Chu Estaing, Clermont-Ferrand
  - Chu Bocage, Dijon
  - Chu de Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Chu Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hopital D'Enfants La Timone, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Chu Nantes, Nantes
  - Chu de Nice, Nice
  - Institut Curie, Paris
  - Chu de Poitiers, Poitiers
  - Chur de Reims, Reims
  - Chu de Rennes, Rennes
  - Chu de Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Hoptial Hautepierre, Strasbourg
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours
  - Chu Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).